CLINICAL TRIAL: NCT05272462
Title: A Phase II Trial of Oral Minoxidil for the Treatment of Recurrent Platinum Resistant Epithelial Ovarian Cancer
Brief Title: Oral Minoxidil for the Treatment of Recurrent Platinum Resistant Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Collaborators: Cures Within Reach (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Margaret Liotta, Associate Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 214787
Record Dates: First submitted 2022-02-09; First posted 2022-03-09 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Platinum Resistant; Epithelial Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Minoxidil

STUDY DESIGN:
Intervention Model Description: This is a non-randomized prospective single-site trial of minoxidil for patients living with recurrent platinum resistant ovarian cancer.
Masking Description: This study is an open-label Phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Participants in this arm will be treated with minoxidil. This treatment will be given daily by mouth.
  Interventions: Drug: Minoxidil

INTERVENTIONS:
Drug: Minoxidil — Minoxidil is an antihypertensive vasodilator medication commonly used for the treatment of high blood pressure and pattern hair loss.
  Other Names: Rogaine

SUMMARY:
The primary purpose of this study is to determine the response rate of patients with recurrent platinum resistant ovarian cancer when treated with oral minoxidil. Secondary objectives include estimating the time to disease progression while on minoxidil and to describe the toxicities of minoxidil when used for patients with recurrent platinum resistant ovarian cancer. An exploratory objective is to evaluate if efficacy of minoxidil is improved in patients that have the Kir6/SUR complex versus those that do not.

DETAILED DESCRIPTION:
Minoxidil is approved by the Food and Drug Administration (FDA) for treatment of hypertension. In previous studies, the sulfonylurea receptor (SUR) subunit controls the selectivity of the pharmacological response to drugs that either inhibit or stimulate the Kir6/SUR channel. Oral minoxidil acts as an activator of the Kir6/SUR2 channel upon selective binding to sulfonylurea receptor 2 (SUR2). Activation of the Kir6.2 potassium channel by minoxidil leads to potassium outflow and calcium entry which produces a cytoplasmic electrical charge that is more negative. This in turn creates an attractive force for calcium to enter the cell. Increased intracellular calcium disrupts mechanisms of cell division by arresting the cell cycle in G2/M phase and this is associated with alteration of the oxidative state, disruption of the mitochondria and activation of the caspase-3-independent cell death pathway.

Evaluation of arrest of tumor growth was evaluated in a previous study. This was done in vitro as well as in vivo by establishing a xenograft model from a Kir6.2/SUR2 positive high grade serous ovarian cancer cell line. In the mice treated with minoxidil, five of the 6 mice had no evidence of measurable disease at necropsy. In contrast, the untreated mice were found to have carcinomatosis and ascites in all 6 mice, demonstrating tumor reduction with minoxidil treatment.

While recurrent ovarian cancer can be treated with a multitude of drugs, the response rates are limited. Treatment options can also be limited secondary to myelosuppression as a result of patients being heavily pretreated. Minoxidil appears to have the advantage of not causing severe myelosuppression which can limit treatment options for patients. Laboratory results provide promising evidence that minoxidil could be used for the treatment of recurrent ovarian cancer.

This study plans to conduct a single center phase II study to evaluate the efficacy and safety of oral minoxidil in the treatment of platinum resistant ovarian cancer. The primary goal is to assess whether treatment with minoxidil will reduce tumor burden in patients with recurrent ovarian cancer and have a minimal toxicity profile.

ELIGIBILITY:
Inclusion Criteria

* Participants must have recurrent platinum resistant ovarian cancer. Histologic documentation of the recurrence is not required.
* Participants must have platinum resistant disease defined as recurrence less than 6 months after initial platinum based treatment.
* Participants must be greater than or equal to 18 years of age.
* Participants must have an Eastern Cooperative Group (ECOG) Performance Status (PS) less than or equal to 2.
* Participants must be able to take oral medications.

Exclusion Criteria

* Participants must not have had chemotherapy or radiotherapy within 4 weeks
* Participants must not be receiving any other investigational agents.
* Participants must not have brain metastases
* Participants must not have allergic reactions to minoxidil
* Participants must not have congestive heart failure
* Participants must not have history of cardiac disease
* Participants must not have uncontrolled hypertension
* Participants must not be on dialysis

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | At the end of Cycle 2 (each cycle is 28 days)
  The ORR is defined as the percentage of participants who experience a complete response (CR), partial response (PR), or stable disease (SD) as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  PFS is defined as the time from receipt of minoxidil to the first documented progression of disease or death due to any cause, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Liotta, DO, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.